CLINICAL TRIAL: NCT05484375
Title: Capecitabine Plus Toripalimab Maintenance Therapy in Metastatic Nasopharyngeal Carcinoma After First-line Gemcitabine/Cisplatin Plus Toripalimab Treatment: a Single Arm, Open Label, Multicenter, Phase II Clinical Study
Brief Title: Capecitabine Plus Toripalimab Maintenance Therapy in Metastatic Nasopharyngeal Carcinoma After First-line Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Hunan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wenjing Yin, attending physician, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-017(FL5)
Record Dates: First submitted 2022-07-30; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; capecitabine; toripalimab; maintenance therapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Capecitabine plus toripalimab maintenance therapy (Experimental): capecitabine and toripalimab were used as maintenance therapy every 3 weeks until toxicity was unacceptable, disease progression, consent withdrawal, or withdrawal was determined by the investigator, or a maximum of 2 years of treatment had been reached.
  Interventions: Drug: Capecitabine plus toripalimab

INTERVENTIONS:
Drug: Capecitabine plus toripalimab — Capecitabine tablet: 650mg/m2, orally, twice a day, d1-d21, every 3 weeks Toripalimab: 240mg, intravenous drip, d1, every 3 weeks

SUMMARY:
to evaluate the efficacy and safety of toripalimab and capecitabine maintenance therapy in patients with metastatic nasopharyngeal carcinoma (NPC) after first-line gemcitabine/cisplatin combined with toripalimab.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy and safety of toripalimab and capecitabine maintenance therapy in patients with metastatic nasopharyngeal carcinoma (NPC) after first-line gemcitabine/cisplatin combined with toripalimab. Patients received a standard dose of toripalimab combined with gemcitabine/cisplatin every 3 weeks (Q3W) for 4-6 cycles. Efficacy was assessed after 4-6 courses of chemotherapy, and patients with PR/CR were enrolled in the clinical trial for maintenance therapy. During maintenance therapy, capecitabine and toripalimab were used as maintenance therapy every 3 weeks until toxicity was unacceptable, disease progression, consent withdrawal, or withdrawal was determined by the investigator, or a maximum of 2 years of treatment had been reached.

ELIGIBILITY:
Inclusion Criteria:

1. Histology confirmed metastatic nasopharyngeal carcinoma following radical treatment（Stage IVb, AJCC/UICC 8th，any T，any N，M1）
2. Patients receiving gemcitabine/cisplatin in combination with terriprizumab received complete response (CR) or partial response (PR) after 4-6 cycles of imaging studies
3. Age ≥18 years and ≤65 years
4. WBC≥4×10^9/L, platelet ≥ 100×10^9/L, hemoglobin ≥ 90g/L and Albumin≥28 g/L
5. With normal liver function test (TBIL#ALT#AST ≤ 2.5×uln) (patients with liver metastasis≤5×uln)
6. With normal renal function test (creatinine ≤ 1.5×uln or CCR ≥ 60ml/min)
7. ECOG score is 0-1
8. At least one measurable lesion according to RECIST v 1.1 (prior to gemcitabine/cisplatin plus toripalimab)
9. Life expectancy is at least 12 weeks
10. Patients sign informed consent forms

Exclusion Criteria:

1. History of severe anaphylaxis to any component of capecitabine or toripalimab
2. Active or untreated central nervous system metastases
3. Patient with necrotic lesions and judged by the investigator to be at risk of excessive bleeding
4. Patients with poorly controlled pleural effusion, pericardial effusion, or ascites requiring frequent drainage. Patients with indwelled catheters are allowed to participate.
5. Patients with poorly controlled or symptomatic hypercalcemia
6. Pregnancy or lactation
7. Malignancies other than nasopharyngeal carcinoma, with negligible risk of metastasis or death and radical outcome expected after treatment, within the 5 years prior to enrollment.
8. Patients who have previously received allogeneic bone marrow transplants or solid organ transplants.
9. History of autoimmune diseases
10. Received systemic immunostimulant therapy (except toripalimab in palliative chemotherapy, including but not limited to interferon or IL-2) within 4 weeks prior to enrollment or during 5 half-lives of the drug.
11. Receive any active vaccine within 4 weeks prior to enrollment
12. Basic medical conditions that the investigator identified as likely to affect significantly drug administration and protocol adherence of the study
13. Active pneumonia
14. Active infections, including tuberculosis, hepatitis B, hepatitis C or HIV.
15. Presence of severe neurological or psychiatric disorders, including dementia and seizures.
16. Peripheral nerves which was graded as≥ 2 according to NCI-CTCAE
17. Major cardiovascular diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival(PFS) | up to 24 month
  The time is defined from the enrolment to progression or death from any cause

SECONDARY OUTCOMES:
overall survival(OS) | up to 24 month
  The time is defined from the enrolment to death from any cause
Objective Response Rate(ORR) | up to 24 month
  The percentage of patients with CR and PR assessed by investigators according to Recist v 1.1
Disease Control Rate (DCR) | up to 24 month
  The proportion of patients who have achieved complete response，partial response and Stable disease assessed by investigators according to Recist v 1.1
Duration of Response (DoR) | up to 24 month
  The time is defined from first documented objective response to radiographic disease progression or death, whichever occurred first, assessed by investigator
Adverse Events (AEs) | up to 24 month
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Yin Wen-Jing, Study Director — Affiliated Cancer Hospital & Institute of Guangzhou Medical University